CLINICAL TRIAL: NCT03890770
Title: An Open-Label, Single-Dose Study to Evaluate the Pharmacokinetics and Safety of BMS-986165 in Participants With Normal Renal Function and Participants With Mild, Moderate, and Severe Renal Impairment and in Participants With End-Stage Renal Disease (ESRD) on Hemodialysis
Brief Title: A Study to Assess the Safety of Experimental Medication BMS986165 in Participants With Normal Kidney Function and Participants With Mild to End-Stage Kidney Disease.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM011-061; 2018-002533-38 (EudraCT Number)
Record Dates: First submitted 2019-03-25; First posted 2019-03-26 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Renal Impairment; Healthy Volunteer
MeSH Terms: conditions — Renal Insufficiency | interventions — deucravacitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Normal renal function (Experimental): Single dose
  Interventions: Drug: BMS-986165
- Mild renal disease (Experimental): Single dose
  Interventions: Drug: BMS-986165
- Moderate renal failure (Experimental): Single dose
  Interventions: Drug: BMS-986165
- Severe renal failure (Experimental): Single dose
  Interventions: Drug: BMS-986165
- End-stage renal disease requiring dialysis (Experimental): Two single doses administered with washout
  Interventions: Drug: BMS-986165

INTERVENTIONS:
Drug: BMS-986165 — Oral administration

SUMMARY:
The purpose of this study is to investigate BMS-986165 in participants with different levels of kidney function.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Participants must be judged to be in good health in the opinion of the investigator OR participant has a stable disease (eg, hypertension, hyperlipidemia, diabetes mellitus, hyperthyreosis) under medical control (ie, no changes in medication within 30 days prior to study drug administration)
* Stable renal impairment, defined as no clinically significant change in disease status, as documented by the participant's most recent eGFR assessment; eGFR must not vary more than 30% from screening to Day -1 to confirm stable renal function, and the renal impairment must be expected by the investigator not to change significantly during the next 3 months
* Body mass index of 18.0 to 38.0 kg/m2, inclusive, and weight ≥50 kg, at screening

Exclusion Criteria:

* Clinically relevant abnormal medical history, abnormal findings on physical examination, vital signs, ECG, or laboratory tests at screening that the investigator judges as likely to interfere with the objectives of the trial or the safety of the participant
* Have a history of cancer (malignancy) with the following exceptions: (1) subjects with adequately treated non-melanomatous skin carcinoma or carcinoma in situ of the cervix may participate in the trial; (2) subjects with other malignancies that have been successfully treated ≥10 years prior to the screening visit where, in the judgment of both the investigator and treating physician, appropriate follow-up has revealed no evidence of recurrence from the time of treatment through the time of the screening visit
* History or clinical evidence of acute or chronic bacterial infection (eg, pneumonia, septicemia) within 3 months prior to screening

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-02-13 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Approximately 9 days
Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration [AUC(0-T)] | Approximately 9 days
Area under the plasma concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] | Approximately 9 days

SECONDARY OUTCOMES:
Incidence of nonserious adverse events (AE), serious adverse events (SAE), and AE leading to discontinuation | Approximately 45 days
Number of clinically significant changes in clinical laboratory values, vital signs, ECGs, and physical examinations | Approximately 45 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (6):
- Orlando Clinical Research Center, Orlando, Florida, United States
- Pharmaceutical Research Associates CZ, s.r.o, Prague, Czechia
- Hungary (2):
  - Szent Imre Egyetemi Oktatokorhaz, Budapest
  - Kenezy Gyula Korhaz es Rendelointezet, Debrecen
- Poland (2):
  - Samodzielny Publiczny Secjalistyczny Szpital Zachodni im. sw. Jana Pawla II, Grodzisk Mazowiecki
  - Specjalistyczne Centrum Medyczne Chirurgii Maloinwazyjnej SCM, Krakow

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm